CLINICAL TRIAL: NCT05886842
Title: Reliability of 30 Seconds Sit-to-stand and Timed Up and Go in Adults With Long Covid
Brief Title: Reliability (Test-retest) of 30 Seconds Sit-to-stand and Timed Up and Go in Adults With Long Covid
Status: Completed | Type: Observational
Sponsor: European University Cyprus (Other)
Collaborators: Eden Resort Wellness Rehabilitation Center (Unknown)
Responsible Party: Principal Investigator, Marina Kloni, Marina Eleni Kloni, BSc, MSc, MA, European University Cyprus
Other Study IDs: Test-Retest
Record Dates: First submitted 2023-04-12; First posted 2023-06-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
Keywords: Test-retest; Reliability; 30 seconds Sit to Stand; Timed up and Go
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Test-retest: A group of 19 patients will be tested using the 30 seconds Sit-to-stand and Timed up and go tests. Each test will be repeated 3 times and the best score will be used. There is going to be 3 days waiting period before the re-tests.
  Interventions: Other: Test-retest

INTERVENTIONS:
Other: Test-retest — Test-retest
  Other Names: Reliability

SUMMARY:
The goal of this study is to test the reliability (with a test-retest process) of 30 seconds Sit to Stand and Timed Up and Go in an adult population with long-covid, hospitalised in a rehabilitation center.

DETAILED DESCRIPTION:
Since December 2019, Covid-19 has affected millions of people worldwide, leaving many of them with symptoms such as fatigue, (muscle) weakness and dyspnoea, even months after their infection (long covid). Rehabilitation centers were established to aid this new group of patients. This study's aim is to test the reliability of 2 outcome measures for patients with long covid. 30 seconds Sit-To-Stand and Timed Up And Go tests are not specific to a disease but they evaluate functionality, mobility and endurance. They are easy to perform in a clinical setting as they do not require specific equipment. The reliability of the above tests has yet to be established in people with long covid.

A sample size of 19 people will be used. A difference in reliability of 0.9 and 0.7 at 80% power and a 5% level of significance using two ratings was set. Based on two testing sessions, an x value of 0.05, and a power of 0.80, a minimal sample size of 19 patients was identified (Karagiannis et al., 2020).

19 patients with long covid from the rehabilitation center will take both tests in a single day and 3 days later they will take the tests again with no physical therapy intervention in between the measurements.

For the statistical analysis, ICC (Intra-class correlation coefficients), SEM (standard error of measurement) and Bland-Altman plot will be used. These tests evaluate test-retest reliability, through the identification of the agreement of patient's scores between the 2 measurements and they evaluate the measurement precision (Savva et al, 2014).

ELIGIBILITY:
Inclusion Criteria:

* Adults who were infected with COVID-19 virus in the last 6 months and were diagnosed with long-covid
* Patients must be willing to give written consent for participation in the study
* Negative rapid test for COVID-19

Exclusion Criteria:

* People under 18 years of age
* Significant cognitive and psychiatric impairments (inability to follow simple commands or give consent)
* Refuse to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of long-covid hospitalised in a rehabilitation center
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Reliability of 30 seconds Sit to stand | Two occasions within approximately three days to establish intra rater reliability
  Test-retest that assess the reliability of 30 seconds Sit to Stand
Reliability of Timed Up and Go | Two occasions within approximately three days to establish intra rater reliability
  Test-retest that assess the reliability of Timed Up and Go

CONTACTS AND LOCATIONS:
Overall Officials: Marina E Kloni, Principal Investigator — European University Cyprus
Locations (1):
- Eden resort wellness rehabilitation, Larnaca, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiredo PHS, Veloso LRS, Lima MMO, Vieira CFD, Alves FL, Lacerda ACR, Lima VP, Rodrigues VGB, Maciel EHB, Costa HS. The reliability and validity of the 30-seconds sit-to-stand test and its capacity for assessment of the functional status of hemodialysis patients. J Bodyw Mov Ther. 2021 Jul;27:157-164. doi: 10.1016/j.jbmt.2021.02.020. Epub 2021 Mar 4. PMID 34391227
- [Background] Hansen H, Beyer N, Frolich A, Godtfredsen N, Bieler T. Intra- and inter-rater reproducibility of the 6-minute walk test and the 30-second sit-to-stand test in patients with severe and very severe COPD. Int J Chron Obstruct Pulmon Dis. 2018 Oct 18;13:3447-3457. doi: 10.2147/COPD.S174248. eCollection 2018. PMID 30425474
- [Background] Ozcan Kahraman B, Ozsoy I, Akdeniz B, Ozpelit E, Sevinc C, Acar S, Savci S. Test-retest reliability and validity of the timed up and go test and 30-second sit to stand test in patients with pulmonary hypertension. Int J Cardiol. 2020 Apr 1;304:159-163. doi: 10.1016/j.ijcard.2020.01.028. Epub 2020 Jan 15. PMID 31980271
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Donner A, Eliasziw M. Sample size requirements for reliability studies. Stat Med. 1987 Jun;6(4):441-8. doi: 10.1002/sim.4780060404. PMID 3629046
- [Background] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853
- [Background] Karagiannis C, Savva C, Korakakis V, Matheou I, Adamide T, Georgiou A, Xanthos T. Test-Retest Reliability of Handgrip Strength in Patients with Chronic Obstructive Pulmonary Disease. COPD. 2020 Oct;17(5):568-574. doi: 10.1080/15412555.2020.1808604. Epub 2020 Aug 19. PMID 32814452
- [Background] Savva C, Giakas G, Efstathiou M, Karagiannis C. Test-retest reliability of handgrip strength measurement using a hydraulic hand dynamometer in patients with cervical radiculopathy. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):206-10. doi: 10.1016/j.jmpt.2014.02.001. Epub 2014 Mar 11. PMID 24630769
- [Background] Shechtman O, Gestewitz L, Kimble C. Reliability and validity of the DynEx dynamometer. J Hand Ther. 2005 Jul-Sep;18(3):339-47. doi: 10.1197/j.jht.2005.04.002. PMID 16059855
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Myles PS, Cui J. Using the Bland-Altman method to measure agreement with repeated measures. Br J Anaesth. 2007 Sep;99(3):309-11. doi: 10.1093/bja/aem214. No abstract available. PMID 17702826
- [Background] Shrout PE. Measurement reliability and agreement in psychiatry. Stat Methods Med Res. 1998 Sep;7(3):301-17. doi: 10.1177/096228029800700306. PMID 9803527